CLINICAL TRIAL: NCT03034941
Title: Short Term Weight Loss With Liraglutide and Metformin Before IVF in Infertile Obese PCOS Patients
Brief Title: Short Term Weight Loss With Liraglutide and Metformin in Infertile Obese PCOS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, professor, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Obesity,PCOS and IVF
Record Dates: First submitted 2017-01-04; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Obesity; PCOS
Keywords: Obesity; PCOS; Infertility; Liraglutide; Metformin; IVF
MeSH Terms: conditions — Obesity; Infertility | interventions — Metformin; Liraglutide; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- metformin group (Active Comparator): Drug: metformin
  Interventions: Drug: Metformin
- COMBI group (Active Comparator): Drug: liraglutide + metformin
  Interventions: Drug: Metformin; Drug: Liraglutide + metformin
- CONTROL group (No Intervention): control group of obese PCOS patients without therapy

INTERVENTIONS:
Drug: Metformin — In the metformin group metformin was initiated at a dose of 500 mg once per day and increased by 500 mg every 3 days up to 1000 mg twice per day per os for 12 weeks
  Other Names: Glucophage tablets
  Arms: COMBI group; metformin group
Drug: Liraglutide + metformin — In the COMBI group the initial dose of metformin was 500 mg for at least 2 wk and gradually increased to a final dose of 1000 mg twice per day. Liraglutide 1.2 mg once per day s.c. was added after first two weeks of monotherapy with metformin.
  Other Names: Victoza 6 mg/ml solution and Glucophage tablets
  Arms: COMBI group

SUMMARY:
The aim of this study was to evaluate the impact of short-term weight reduction achieved with 12-week intervention with metformin alone or in combination with liraglutide on oocyte maturity and embryo quality in infertile obese PCOS population.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common cause of anovulatory infertility, in particular when PCOS is linked to obesity. Obese PCOS has poor IVF outcomes associated with impaired oocyte and embryo parameters and morphology. The purpose of this pilot prospective study was to investigate the effect of the antiobesity medical therapy (combination of metformin and liraglutide (COMBI)) on short time weight loss in the specific infertile obese PCOS population. Additionally, we analyzed eventual impact of the short term weight loss 5% or more before IVF on oocyte maturity and embryo quality in infertile obese PCOS population.

ELIGIBILITY:
Inclusion Criteria:

* polycystic ovary syndrome (rotterdam criteria)
* BMI of 30 kg/m² or higher
* Infertility for IVF with normal male sperm

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus
* history of carcinoma
* Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
* personal or family history of multiple endocrine neoplasia 2
* significant cardiovascular, kidney or hepatic disease
* the use of medications known or suspected to affect reproductive or metabolic functions
* the use of statins, within 90 days prior to study entry

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The main outcome was change in BMI | Patient's BMI was measured at the beginning and every four weeks during 12 weeks of clinical trial.

SECONDARY OUTCOMES:
Impact of the short term weight loss 5% or more before IVF on oocyte maturity in infertile obese PCOS population. | patients were introduced to IVF one month after completed weight loss therapy
Impact of the short term weight loss 5% or more before IVF on oocyte number of blastocysts in infertile obese PCOS population. | patients were introduced to IVF one month after completed weight loss therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eda Vrtacnik Bokal, professor, Study Chair — University Medical Centre Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Data are going to be available for other researchers if needed after the evaluation of this study.

REFERENCES:
- [Background] Jensterle Sever M, Kocjan T, Pfeifer M, Kravos NA, Janez A. Short-term combined treatment with liraglutide and metformin leads to significant weight loss in obese women with polycystic ovary syndrome and previous poor response to metformin. Eur J Endocrinol. 2014 Feb 7;170(3):451-9. doi: 10.1530/EJE-13-0797. Print 2014 Mar. PMID 24362411
- [Background] Jungheim ES, Lanzendorf SE, Odem RR, Moley KH, Chang AS, Ratts VS. Morbid obesity is associated with lower clinical pregnancy rates after in vitro fertilization in women with polycystic ovary syndrome. Fertil Steril. 2009 Jul;92(1):256-61. doi: 10.1016/j.fertnstert.2008.04.063. Epub 2008 Aug 9. PMID 18692801
- [Background] Depalo R, Garruti G, Totaro I, Panzarino M, Vacca MP, Giorgino F, Selvaggi LE. Oocyte morphological abnormalities in overweight women undergoing in vitro fertilization cycles. Gynecol Endocrinol. 2011 Nov;27(11):880-4. doi: 10.3109/09513590.2011.569600. Epub 2011 Apr 18. PMID 21500991